CLINICAL TRIAL: NCT04086290
Title: Oligomet-DK. National Danish Protocol. Surgery+ SBRT for M1 Prostate Cancer Patients
Brief Title: National Danish Protocol. Surgery+ SBRT for M1 Prostate Cancer Patients
Acronym: Oligomet_DK
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Peter Busch Østergren (Other)
Responsible Party: Sponsor-Investigator, Peter Busch Østergren, Principal Investigator, Herlev Hospital
Organization: Herlev Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Oligomet_DK
Record Dates: First submitted 2019-09-02; First posted 2019-09-11 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Prostate Cancer Metastatic
Keywords: radiotherapy; prostatectomy; androgen deprivation therapy
MeSH Terms: interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RARP + SBRT + ADT (Experimental): Radical prostatectomy + extended pelvic lymph node dissection according to EAU guidelines followed by stereotactic body radiotherapy to osseous lesions with six month of neo-adjuvant/concomitant medical castration therapy using a gonadotropin-releasing hormone antagonist or agonist.
  Interventions: Procedure: RARP; Radiation: SBRT; Drug: ADT

INTERVENTIONS:
Procedure: RARP — Radical prostatectomy + extended pelvic lymph node dissection
  Other Names: Robot assisted Radical Prostatectomy
Radiation: SBRT — Stereotactic body radiotherapy to osseous lesions
  Other Names: Stereotactic body radiotherapy
Drug: ADT — six month of neo-adjuvant/concomitant medical castration therapy using a gonadotropin-releasing hormone antagonist or agonist.
  Other Names: Androgen deprivation therpay

SUMMARY:
A prospective, open label phase 2 clinical trial assessing safety, complications and feasibility of radical prostatectomy (RARP) plus local stereotactic body radiotherapy (SBRT) to bone metastases in combination with short-term medical castration to a select population of prostate cancer patients with oligometastatic disease.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older and willing and able to provide informed consent;
2. Stage cT1 ≤ cT3b, Clinical resectable
3. Gleason score ≥ 6
4. M1

   1. ≤ 3 bone metastases localized to the spine, pelvis or humeral/femoral bones as evaluated by 68Ga-PSMA PET/CT and magnetic resonance imaging (MRi)
   2. Absence of PSMA uptake in retroperitoneal lymph nodes, (outside the anatomical region of extended pelvic lymph node dissection as described in the European Association of Urology (EAU) guidelines.
   3. No visceral metastasis
   4. Metastases suitable for stereotactic body radiotherapy
   5. Non symptomatic bone lesions
5. Eligible for surgery

Exclusion Criteria:

1. Prior curative intended treatment for prostate cancer
2. Prior androgen deprivation therapy (ADT)
3. History of another invasive cancer within 3 years of screening, with the exception of fully treated cancers with a remote probability of recurrence. The medical monitor and investigator must agree that the possibility of recurrence is remote for exceptions.
4. Eastern Cooperative Oncology Group (ECOG) Performance Status > 1
5. Evaluated not able to fulfil the study protocol.
6. Contraindications against MRI

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-10-10 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Proportion of men with Grade ≥ 3 adverse events the first year | 1 year
  Proportion of men with Grade ≥ 3 adverse events the first year

SECONDARY OUTCOMES:
Proportion of men achieving prostatic specific antigen (PSA) < 0.1 ng/ml | 1 year
  Proportion of men achieving prostatic specific antigen (PSA) < 0.1 ng/ml
Feasibility of radical prostatectomy in the oligometastatic setting | 1 year
  Feasibility of radical prostatectomy in the oligometastatic setting measured as number of patients who successfully undergo radical prostatectomy with pelvic lymphnode disection and 30 days (post-operative) morbidity according to the Clavian Dindo Classification.

OTHER OUTCOMES:
Time to castrate resistance (TCR) | 5 yrs
  Time to castrate resistance (TCR) measured from the primary initiation of ADT to Castrate Resistant Prostate Cancer (CRPC) defined as: Three consecutive rises in PSA one week apart resulting in two 50% increases over the nadir, with PSA > 1 ng/mL or the appearance of two or more new bone lesions on bone scan or enlargement of a soft tissue lesion using RECIST. At the same time serum testosterone is <50ng/dL (<1.70 nnmol/L).
Quality of life (FACT-P-DK) | 5 yrs
  Changes in Quality of life assessed by the questionaire FACT-P-DK and calculated using the FACT-P Scoring Guidelines (Version 4). The following scores will be evaluated:
  1. FACT-P Trial Outcome Index (TOI). Score range: 0-104 (The higher score the better). Combines the subscales "Physical well-being", "Functional Well-being" and "Prostate Cancer Subscale"
  2. FACT-G total score. Score range: 0-108 (the higher score the better QoL). Combines the subscales: "Physical well-being", "Social well-being", "Emotional well-being" and "Functional well-being".
  3. FACT-P total score. Score range: 0-156 (the higher score the better QoL). Combines the subscales: "Physical well-being", "Social well-being", "Emotional well-being", "Prostate Cancer Subscale" and "Functional well-being".
Number of participants with Interventions on lower or upper urinary tract | 5 yrs
  Number of participants undergoing with interventions on lower or upper urinary tract, i.e.:
  * Bladder catheter
  * Ureteric stent
  * Nephrostomy
  * Transurethral resection of the prostate (TURP) or related procedure

CONTACTS AND LOCATIONS:
Overall Officials: Peter B Østergren, MD, Principal Investigator — Herlev and Gentofte Hospital
Locations (1):
- Herlev and Gentofte Hospital, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No